CLINICAL TRIAL: NCT06254950
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled, Double-Blind Induction Study to Evaluate the Efficacy and Safety of Oral TAK-279 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study on the Safety of TAK-279 and Whether it Can Reduce Inflammation in the Bowel of Participants With Moderately to Severely Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-279-UC-2001; 2023-506769-67-00 (EU CTIS Number: Abbreviated EU CT Number); jRCT2031240228 (Registry Identifier: jRCT)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Drug Therapy; Latitude UC, Latitude Research Program
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TAK-279 Dose 1 (Experimental): TAK-279, capsules, orally at Dose 1 up to Week 12 followed by either Dose 1 or Dose 2 up to week 52 based on the response.
  Interventions: Drug: TAK-279
- TAK-279 Dose 2 (Experimental): TAK-279, capsules, orally at Dose 2 up to Week 12 followed by either Dose 1 or Dose 2 up to week 52 based on the response.
  Interventions: Drug: TAK-279
- Placebo (Placebo Comparator): TAK-279 matching placebo capsules, orally, for 12 weeks followed by TAK-279 capsules, orally either Dose 1 or Dose 2 up to Week 52 based on the response.
  Interventions: Drug: TAK-279; Drug: Placebo

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsules.
  Other Names: Zasocitinib
Drug: Placebo — TAK-279 placebo-matching capsules.
  Arms: Placebo

SUMMARY:
The main aim of this study is to learn if TAK-279 reduces bowel inflammation and symptoms compared to placebo. Another aim is to compare any medical problems that participants have when they take TAK-279 or placebo and how well the participants tolerate any problems.

The participants will take capsules of either TAK-279 or placebo for up to 3 months (12 weeks). Then all the participants will receive TAK-279 for the rest of the treatment part of the study (1 year or 52 weeks).

During the study, participants will visit their study clinic several times.

DETAILED DESCRIPTION:
Study TAK-279-UC-2001 is a multicenter, randomized, placebo-controlled, study with a 12-week double-blinded induction treatment period, a 40-week open-label treatment period (52 total weeks of treatment), and a 4-week safety follow-up period.

An approximate total of eligible 207 participants will be randomized to one of the three treatment groups -

1. TAK-279 Dose 1
2. TAK-279 Dose 2
3. Placebo

The maximum study duration per participant is approximately 60 weeks, including up to 30 days for the screening period, a 12-week randomized and double-blinded induction treatment period, a 40-week open-label treatment period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years old with diagnosis of UC for at least 30 days. In South Korea, the age requirement for adult participants is ≥19 years of age.
2. Confirmed diagnosis of moderately to severely active UC assessed by mMS and ES.
3. Participants with a history of inadequate response to, loss of response to, or intolerance to one or more of conventional, biologic or advance therapies for UC.
4. Participants must meet the contraception recommendations.

Exclusion Criteria:

1. Participants with indeterminate/unclassified inflammatory bowel disease (IBD), microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, diverticular disease associated with colitis, and/or clinical/histologic findings suggestive of Crohn's disease (CD).
2. Participants with complications of UC such as strictures, stenoses, fistulas, short gut syndrome, or any other manifestation that might require surgery during the study.
3. Participants with a current ileostomy or colostomy. Participants who had a J-pouch are excluded, as a J-pouch could result in a stoma.
4. Participants who have failed 3 or more classes of advanced therapies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission at Week 12 Based on Modified Mayo Score (mMS) | Week 12
  The mMS is a composite score of 3 assessments consisting of stool frequency (SF), rectal bleeding (RB), and endoscopic score (ES). Each component subscore ranges from 0 to 3 and total score range of the mMS is from 0 to 9, with higher scores indicating more severe disease. Clinical remission is defined an mMS of ≤2 with SF subscore ≤ 1, RB subscore = 0, and ES ≤ 1 (score of 1 modified to exclude friability).

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response at Week 12 Based on Modified Mayo Score (mMS) | Baseline, Week 12
  Clinical response defined as reduction from baseline in mMS of ≥2 points and ≥30% from baseline and a decrease from baseline in the RB subscore of ≥1 point or an absolute RB subscore of ≤1 point at Week 12.
Percentage of Participants Achieving Symptomatic Remission at Week 12 | Week 12
  Symptomatic remission is defined as a RB subscore of 0 and SF subscore of ≤1.
Percentage of Participants Achieving Endoscopic Improvement at Week 12 | Week 12
  Endoscopic improvement defined as a modified Mayo ES of ≤1 (score of 1 modified to exclude friability).
Percentage of Participants Achieving Endoscopic Remission at Week 12 | Week 12
  Endoscopic remission defined as a modified Mayo ES of 0.
Percentage of Participants With no Bowel Urgency at Week 12 | Week 12
  Bowel urgency measured by the bowel urgency electronic diary (eDiary) item at Week 12.
Percentage of Participants With no Abdominal Pain at Week 12 | Week 12
  Abdominal pain measured by abdominal pain eDiary item at Week 12.
Percentage of Participants With Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score ≥170 at Week 12 | Week 12
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel function (10 items), emotional status (12 items), systemic symptoms (5 items), and social function (5 items). The total score ranges from 32 to 224, with higher scores representing better quality of life.
Change From Baseline in Disease-Specific Health-related Quality of Life (HRQoL) as Measured by IBDQ Total Score at Week 12 | Baseline and Week 12
  The IBDQ is a 32-item questionnaire that measures 4 dimensions: bowel function (10 items), emotional status (12 items), systemic symptoms (5 items), and social function (5 items). The total score ranges from 32 to 224, with higher scores representing better quality of life.
Change From Baseline in Fatigue as Measured by the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Score at Week 12 | Baseline and Week 12
  The FACIT-Fatigue is a reliable and valid instrument for measuring fatigue. The responses to the 13 items on the FACIT-Fatigue questionnaire are each measured on a 5-point Likert scale, where 0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit and 4=Very much. The total score ranges from 0 to 52. High scores represent less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (140):
- United States (16):
  - GastroIntestinal BioSciences, Los Angeles, California
  - United Medical Doctors, Murrieta, California
  - West Central Gastroenterology, LLP, d/b/a/ Gastro Florida, Clearwater, Florida
  - Auzmer Research, Lakeland, Florida
  - GI PROS, Inc., Naples, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida
  - Emory University Hospital, The Emory Clinic, Atlanta, Georgia
  - Atlanta Center For Gastroenterology, P.C., Decatur, Georgia
  - University Of Louisville, Louisville, Kentucky
  - Woodholme Gastroenterology Associates, Glen Burnie, Maryland
  - Las Vegas Medical Research, Las Vegas, Nevada
  - University Gastroenterology, Providence, Rhode Island
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Novel Research, LLC, Bellaire, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - University of Washington Medical Center, Seattle, Washington
- Australia (9):
  - Concord Repatriation General Hospital, Sydney, New South Wales
  - Mater Cancer Care Centre-Mater Health Services, South Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Western Health/Footscray Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital Lung Institute Of Western Australia, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Harry Perkins Medical Research Institute Fiona Stanley Hospital, Murdoch
- Belgium (2):
  - Hopital Universitaire de Bruxelles/ Academisch Ziekenhuis Burssel, Brussels, Anderlecht / Region Capitale de Bruxelles/ Brussel
  - Universitair Ziekenhuis Leuven, Leuven
- Bulgaria (6):
  - UMBAL Kaspela, Plovdiv
  - Pecs University Clinical Center Mohacs Hospital, Sofia
  - Acibadem City clinic Tokuda hospital, Sofia
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia
  - University Hospital Tsaritsa Yoanna - Isul (University Hospital Queen Giovanna), Sofia
  - University Hospital City Clinic Cancer Center, Sofia
- Canada (6):
  - Heritage Medical Research Clinic - University Of Calgary, Calgary, Alberta
  - Fraser Clinical Trials, New Westminster, British Columbia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Center, Montreal, Quebec
- China (10):
  - Chongqing General Hospital, Chongqing, Chongqing Sheng
  - Sun Yat-sen University - The Sixth Affiliated Hospital (Guangdong Gastrointestinal Hospital), Guangzhou, Guangdong
  - Wuhan University - Renmin Hospital (Hubei General Hospital), Chongqing, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Changzhou, Changzhou, Jiangsu
  - China Medical University (CMU) - Shengjing Hospital (The Second Affiliated Hospital) - Huaxiang Campus, Shenyang, Liaoning
  - Renji hospital shanghai jiao tong university school of medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Zhejiang University School of Medicine - Sir Run Run Shaw Hospital (SRRSH), Hangzhou
  - Shanghai Pudong New District Zhoupu Hospital, Shanghai
- Czechia (11):
  - NH Hospital, Hořovice, Central Bohemia
  - SurGal Clinic SRO, Brno
  - Vojenska Nemocnice Brno, Brno
  - University Hospital Brno, Brno
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - EndoArt, Ostrava
  - Fakultni Nemocnice Ostrava (FNO), Ostrava-Poruba
  - Gastromedic s.r.o, Pardubice
  - Endohope Clinic, Prague
  - Axon Clinical s.r.o., Prague
  - Masaryk Hospital, Ústí nad Labem
- Denmark (6):
  - Odense Universitetshospital (OUH) (Odense University Hospital), Odense, Region Syddanmark
  - Aalborg Hospital, Aalborg
  - Sydvestjysk Region/Esbjerg Hospital, Esbjerg
  - Hillerod Hospital, Hilleroed Sygehus, Hillerød
  - Hvidovre Hospital Medicinsk Gastroenterologisk Afdeling, Hvidovre
  - Region Sjaelland Sygehus Nord, Koge Sygehus, Køge
- France (4):
  - CHU De Clermont Ferrand - Hopital Estaing, Clermont-Ferrand
  - Hopital l'Archet 2, Nice
  - Hopital Nord Chu Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Regional Universitaire de Nancy Hopital Brabois, Vandœuvre-lès-Nancy
- Germany (7):
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Hamburger Forschungsinstitut Fuer Chronisch Entzuendliche Darmerkrankungen (HaFCED e.K.), Hamburg
  - Praxis fur Gastroenterologie, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, UKSH-Campus Kiel, Kiel
  - St. Marien- und St. Annastiftskrankenhaus, Ludwigshafen
  - Universitaetsklinikum Tuebingen, Tübingen
  - University Hospital Of Ulm, Universitatsklinikum Ulm, Ulm
- Greece (5):
  - University General Hospital of Patras, Pátrai, Achaia
  - Evaggelismos Hospital (Evangelismos Hospital)-University of Athens, Athens, Attica
  - University Hospital of Heraklion, Heraklion, Crete
  - Sotiria General Hospital of Athens, Athens
  - G.N.A. Gennimatas, Athens
- Hungary (5):
  - Clinexpert, Budapest
  - Semmelweis Egyetem, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Mohacsi Korhaz, Mohács
  - Javorszky Odon Korhaz, Vác
- Israel (4):
  - Assuta Ashdod University Hospital, Ashdod
  - Soroka Mc, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
  - The Chaim Sheba Medical Center - The Edmond and Lily Safra Children's Hospital, Ramat Gan
- Italy (5):
  - IRCCS A.O.U. Policlinico S. Orsola - Malpighi, Bologna
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele Hospital, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - Azienda Ospedaliera San Camillo Forlanini, Rome
  - IRCCS Istituto clinico humanitas - Humanitas Mirasole spa, Rozzano
- Japan (8):
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kansai Medical University Hospital, Hirakata, Osaka
  - The jikei University Hospital, Minato, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - Saga University Hospital, Saga
- Norway (2):
  - Akershus University Hospital, Lorenskog, Akershus
  - Oslo Univeristy Hospital Ulleval Hospital, Oslo
- Poland (12):
  - Centrum Medyczne Melita Medical, Wroclaw, Dolnolskie
  - Gastromed Kopon, Zmudzinski i Wspolnicy Sp.j. Specjalistyczne Centrum Gastrologii i Endoskopii Specjalistyczne Gabinety Lekarskie, Torun, Kujawsko-pomo
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - PlanetMed Sp. z o.o., Wroclaw, Lower Silesian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA, Warsaw, Masovian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - Oddzial Kliniczny Gastroenterologii Ogolnej i Onkologicznej SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Medrise sp. z o.o, Lublin
  - Centrum Medyczne MedykSp. z o.o. Sp. K., Rzeszów
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - H-T. Centrum Medyczne Sp. z o.o. Sp.k., Tychy
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Romania (5):
  - Policlinica Algomed: Centrul De Gastroenterologie Dr. Goldis, Timișoara, Jud Timis
  - Clinical Hospital Colentina-Spitalul Clinic Colentina, Bucharest
  - Spitalul de Oncologie Monza - Soseaua Gheorghe Ionescu Sisesti, Bucharest
  - Delta Health Care, Bucharest
  - Spital Clinic Dr I Cantacuzino, Bucharest
- Slovakia (5):
  - Fakultna nemocnica F. D. Roosevelta, Banská Bystrica
  - Cliniq s. r. o., Bratislava
  - Endomed, Košice
  - Fakultna Nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Accout Center, s.r.o.- Gastroenterologicka ambulancia, Šahy
- South Korea (5):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inje University Haeundae Paik Hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center (AMC), Seoul
  - Samsung Medical Center, Seoul
- Taiwan (3):
  - Changhua Christian Hospital (CCH), Changhua, Changhua County
  - National Taiwan University Hospital (NTUH), Taipei, Zhongzheng District
  - China Medical University Hospital, Taichung
- United Kingdom (4):
  - Clinical Research Centre - Barts Health NHS Trust, London, E1 2at
  - South Eastern Health and Social Care Trust - The Ulster Hospital, Belfast
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - St Thomas' Hospital - Guy's & St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/3918b50bd98446ef?idFilter=%5B%22TAK-279-UC-2001%22%5D